CLINICAL TRIAL: NCT07112092
Title: Therapeutic Play and Music Therapy in Dental Anxiety Management: A Randomised Clinical Trial
Brief Title: Therapeutic Play and Music Therapy in Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, Assoc. Prof., Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/279
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Behavior Management; Music Therapy
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: (n=42) control (Tell-Show-Do) group (Active Comparator): The treatment procedure and the exact steps were explained to the child verbally, after which all the tools and equipment required for the treatment were shown to the child before the extraction was performed.
  Interventions: Behavioral: Tell-Show-Do
- Group 2: (n=42) tell-show-do with music therapy application group (Experimental): The planned tooth extraction had been explained to the children using the Tell-Show-Do (TSD) technique, and each child had been asked to select a preferred song. During the procedure, the selected songs were played on a screen mounted in the dental unit. The duration of the therapy had been standardized to 10 minutes in order to relax the children's physiological and psychological state.
  Interventions: Behavioral: Music Therapy
- Group 3: (n=42) tell-show-do with therapeutic play therapy application group (Experimental): For the TSD and therapeutic play therapy groups, a play therapy-certified researcher demonstrated the procedure on a model using a plush Pink Panther toy (Youya Dental Supply Store, China) and a toy dentist set (Heroes Toys, Turkey). Children were allotted 10 minutes to roleplay the procedure, interact with the toys to facilitate emotional expression related to the procedure, and ask any questions.
  Interventions: Behavioral: Therapeutic Play Therapy

INTERVENTIONS:
Behavioral: Tell-Show-Do — Standard behavioral management technique where the dental procedure is explained to the child, demonstrated, and then performed.
  Arms: Group 1: (n=42) control (Tell-Show-Do) group
Behavioral: Music Therapy — Participants listen to calming music during the dental extraction procedure to reduce anxiety and pain perception.
  Arms: Group 2: (n=42) tell-show-do with music therapy application group
Behavioral: Therapeutic Play Therapy — Use of structured play activities designed to reduce dental anxiety and improve cooperation during tooth extraction.
  Arms: Group 3: (n=42) tell-show-do with therapeutic play therapy application group

SUMMARY:
This study aims to evaluate the effects of therapeutic play and music therapy on dental anxiety and pain levels in pediatric patients undergoing tooth extraction.

DETAILED DESCRIPTION:
A total of 126 children aged 6-8 years who required maxillary molar extraction were randomly assigned to three groups (n=42): a control group (Tell-Show-Do), a music therapy group, and a therapeutic play group. Vital signs, including heart rate, blood pressure, oxygen saturation, and body temperature, were recorded. The Modified Child Dental Anxiety Scale - faces version (MCDASf) and the Facial Image Scale (FIS) were used to assess anxiety levels before and after the extraction. Following the extraction, the Wong-Baker Faces Pain Rating Scale (WBFPRS) was used to evaluate pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-8 years
* Scored 3 (positive) or 4 (definitely positive) on the Frankl Behavior Scale
* Systemically healthy
* Had no hearing impairments or allergies
* Had an indication for extraction of any primary maxillary molars (54, 55, 64, 65)
* Whose parents provided informed consent for participation

Exclusion Criteria:

* Had systemic diseases or allergies
* Scored 1 (definitely negative) or 2 (negative) on the Frankl Behavior Scale
* Were undergoing psychological or psychiatric treatment
* Had physical or mental disabilities

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) and diastolic blood pressure (DBP) measurement | 1 month
  The primary outcomes of this study were assessed through physiological measurements (blood pressure).
  Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were recorded at multiple time points during the procedure: before the procedure, after the administration of local anesthesia, after pulpotomy, and at the end of the procedure.
  Each patient had rested for 15 minutes prior to the blood pressure measurement. Measurements were taken from the right wrist with the child in an upright position using an automatic wrist blood pressure device (Wohler, Türkiye).
  Systolic (SBP) and diastolic blood pressure (DBP) values, expressed in centimeters of mercury (cmHg), were recorded.
Heart rate (HR) measurement | 1 month
  The primary outcomes of this study were assessed through physiological measurements (heart rate).
  Heart rate (HR) was measured while the child was in a seated position using a finger-type portable pulse oximeter (Oncomed, USA) attached to the child's right finger. HR values displayed on the digital monitor were recorded as beats per minute.
Hemoglobin oxygen saturation (SpO₂) measurement | 1 month
  The primary outcomes of this study were assessed through physiological measurements (hemoglobin oxygen saturation).
  Hemoglobin oxygen saturation (SpO₂) was measured while the child was in a seated position using a finger-type portable pulse oximeter (Oncomed, USA) attached to the child's right finger. SpO₂ values displayed on the digital monitor were recorded as a percentage.
The Faces Version of the Modified Child Dental Anxiety Scale (MCDASf) measurement | 1 month
  The primary outcomes of this study were assessed through psychometric measurements (The Faces Version of the Modified Child Dental Anxiety Scale).
  The Faces Version of the Modified Child Dental Anxiety Scale (MCDASf) was used to measure the level of anxiety experienced by the children throughout the procedure.
  This scale included five possible responses consisting of smiling or sad faces, appropriate for each answer given by the child. A happy face corresponded to 1 point, whereas a very sad face corresponded to 5 points.
  After the dental treatment, the children in all three groups were asked the questions. The scores corresponding to the selected facial expressions were chosen by the children and recorded by the pediatric dentist.
  The total score was calculated with a minimum of 8 and a maximum of 40, with higher scores indicating greater levels of anxiety.
The Wong-Baker Faces Pain Rating Scale (WBFPRS) measurement | 1 month
  The primary outcomes of this study were assessed through evaluation of dental pain perception (The Wong-Baker Faces Pain Rating Scale).
  The Wong-Baker Faces Pain Rating Scale (WBFPRS) was utilized to assess the pain intensity as reported by the children during the dental treatment.
  The WBFPRS included six facial expressions ranging from a smiling face to a crying face.
  These expressions were explained to the children, who were then asked to choose the face that best reflected the level of pain they felt during the treatment. A smiling face corresponded to 0 points (no pain), whereas a crying face corresponded to 10 points (very severe pain). After physiological and psychometric measurements were recorded, the pediatric dentist used the WBFPRS score to evaluate the children's pain perception. The scoring was recorded by the same pediatric dentist.
  Higher dental anxiety was associated with an increasing score.
The Facial Image Scale (FIS) measurement | 1 month
  The Facial Image Scale (FIS) was specifically designed for children aged 4-12 years and enabled individuals with limited verbal communication skills to express their emotions through facial expressions. The scale consisted of five different facial expressions, rated from 1 (very happy) to 5 (very sad). Children were asked to select the facial expression that best represented their feelings, and their responses were recorded. The FIS was administered both pre-procedure and post-procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No